CLINICAL TRIAL: NCT05145998
Title: Metabolic Effects of Pulse Consumption on Biomarkers in Adults With Type 2 Diabetes Mellitus or Metabolic Syndrome
Brief Title: Metabolic Effects of Pulse Consumption on Biomarkers in Adults With Type 2 Diabetes or Met Syn
Acronym: PGRIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Collaborators: USA Dry Pea & Lentil Council (Unknown)
Responsible Party: Principal Investigator, Donna Winham, Assistant Professor, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17-191
Record Dates: First submitted 2020-01-16; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Type2 Diabetes Mellitus; Metabolic Syndrome
Keywords: Glycemic response; Glucose; Type 2 diabetes; Legumes; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2 | interventions — Glucola

STUDY DESIGN:
Intervention Model Description: 5 x 5 crossover study with 4 treatments and one control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control - Glucola (Active Comparator): Glucola control beverage
  Interventions: Dietary Supplement: Glucola
- Whole peas (Experimental): Whole cooked peas in a 50 gram carbohydrate meal dose
  Interventions: Dietary Supplement: Whole pea meal
- Pea Flour (Experimental): Pea flour in a 50 gram carbohydrate meal dose
  Interventions: Dietary Supplement: Pea flour meal
- Whole lentils (Experimental): Whole cooked lentils in a 50 gram carbohydrate meal dose
  Interventions: Dietary Supplement: Whole lentils
- Lentil flour (Experimental): Lentil flour in a 50 gram carbohydrate meal dose
  Interventions: Dietary Supplement: Lentil flour

INTERVENTIONS:
Dietary Supplement: Glucola — 50 grams of Glucola sugar beverage
  Arms: Control - Glucola
Dietary Supplement: Whole pea meal — Whole cooked peas with spaghetti sauce and a slice of bread.
  Arms: Whole peas
Dietary Supplement: Pea flour meal — Pea flour with spaghetti sauce and a slice of bread.
  Arms: Pea Flour
Dietary Supplement: Whole lentils — Whole cooked lentils with spaghetti sauce and a slice of bread.
  Arms: Whole lentils
Dietary Supplement: Lentil flour — Lentil flour with spaghetti sauce and a slice of bread.
  Arms: Lentil flour

SUMMARY:
The purpose of this study is to determine glycemic response of four different meals containing either whole green peas, whole lentils, powdered green peas, or powdered lentils in comparison to Glucola. Participants are adults with type 2 diabetes mellitus or metabolic syndrome.

DETAILED DESCRIPTION:
The 5 test treatments (Glucola, whole green peas, green pea flour, whole lentils, and lentil flour) will be administered randomly over five weeks. The test Participants will be required to consume the entire test treatment meal in 12 minutes while being observed. Venous blood samples will be collected for blood glucose and insulin levels at time 0 (fasting) and at 30, 60, 90, 120, and 180 minutes post-treatment (timing of the post-treatment blood draws started at time 0 [post-treatment], which is when the participant finishes consuming the treatment meal). During the first visit blood was drawn for a lipid panel and HbA1C values. Thyroid stimulating hormone (TSH) and complete blood count (CBC) values were analyzed during the second visit, and vitamin D levels analyzed during the final visit. Blood analysis was completed by a reputable biomarker diagnostics laboratory, Quest Diagnostics. Anthropometric measures such as weight, height, waist circumference, and blood pressure were collected at screening and at the start of each test day. Thirteen hours before testing, participants consumed a standardized frozen meal to reduce the potential variation in glycemic responses on test day due to varying pre-evening dietary intakes. This control meal was selected by each participant before the start of the study. Each participant was provided the same frozen meal every time, since the subjects serve as their own controls. The day before test day, participants completed a 24 hour food recall, satiety, and gastrointestinal questionnaires. The morning of each test day participants completed the International Physical Activity Questionnaire (IPAQ), satiety, and gastrointestinal questionnaires. Test meal and blood glucose results at the 5 test points were entered into SPSS statistical software (V. 25) for data cleaning and analysis. Physical activity and the 24 hour dietary recall data were used to classify individuals on activity and dietary quality. Satiety responses were compared against each of the 5 test meals for each participant as well as the gastrointestinal responses using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Age 24-70 years
* BMI between 22-40
* Medical diagnosis of type 2 diabetes
* HbA1C <10%)
* OR have 3+ indicators of metabolic syndrome (high triglycerides, low HDL-cholesterol, high blood pressure) plus prediabetes HbA1c.

Exclusion Criteria:

* Uncontrolled hypertension or other health issues, e.g., gastrointestinal disease
* Weight changes of >10% of participants body weight within a 6 month period
* Pregnant or breastfeeding
* Allergy to peas, lentils, tomatoes, gluten, or latex
* HgbA1c level of >10% at screening
* Unwillingness or inability to follow study protocol.

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Change in baseline blood glucose over 3 hours (glycemic response) | Time 0 (fasting) then every 30 minutes for 3 hours
  Venous blood samples were collected via venous catheter. Whole blood samples were analyzed for glucose content and insulin at Quest Diagnostics.

SECONDARY OUTCOMES:
Change in gastrointestinal symptoms | 3 hours postprandial, and 12 hours postprandial
  Gastrointestinal concerns and changes were noted on a descriptive questionnaire
Change in satiety sensation | Time 0 (fasting) then every 30 minutes for 3 hours
  Satiety level measured using a visual analog scale (0-100) every 30 minutes postprandially. A higher score indicates greater satiety.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Winham, DrPH, Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Food Science and Human Nutrition Department, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: No